CLINICAL TRIAL: NCT02251418
Title: Extracorporeal Shockwave Therapy (ESWT) of Chronic Diabetic Foot Ulcers
Brief Title: Shockwave Therapy of Chronic Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Sune Moeller Jeppesen, Medical student, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-ESWTULCER
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Diabetic Foot Ulcer
Keywords: Foot ulcer, diabetic; ESWT (Extracorporeal Shockwave Therapy); Endocrinology; Dermatology; Wound healing; Ischemia; Neovascularization, Physiologic; Pain management
MeSH Terms: conditions — Diabetic Foot; Ischemia; Neovascularization, Pathologic; Agnosia | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Extracorporeal shockwave therapy (Experimental): 6 times extracorporeal shockwave therapy in 3 weeks. This arm also receives standard care treatment.
  Interventions: Device: Extracorporeal shockwave therapy
- Control (No Intervention): Standard care treatment

INTERVENTIONS:
Device: Extracorporeal shockwave therapy
  Other Names: STORZ DUOLITH SD1 T-top shockwave device
  Arms: Extracorporeal shockwave therapy

SUMMARY:
Introduction:

Foot ulcers are a feared complication among diabetic patients. The ulcers can cause pain, discomfort and reduced quality of life. The development of foot ulcers places the patients at a risk of amputation. In the Danish Health Care System a substantial effort is done to prevent and treat diabetic foot ulcers. A constant research of how to treat these wounds is ongoing. The goal is to optimize wound healing and prevent amputations.

Extracorporeal shockwave therapy (ESWT) involves the use of a device that generates low-energy shockwaves through a headpiece, which is placed on the skin of the patient. A small amount of energy will be deposited in the tissue when shockwaves are applied. This stimulates the cells to produce substances that generate new vessels. No side effects to ESWT have been shown.

Purpose:

The investigators want to test whether shockwave therapy can improve wound healing among diabetic patients with foot ulcers.

Hypothesis:

The investigators hypothesize that shockwave therapy accelerates ulcer healing, increases blood flow, reduces pain, and has no side effects.

Method:

Patients who are interested in participation will be included in the study and divided by randomization into two groups of equal size. The first group is treated with ESWT in combination with regular guideline treatment. The second group is set up as control group and will only receive regular guideline treatment. The participants are examined in different ways to evaluate whether ESWT helps the healing of foot ulcers. The investigators want to measure tissue oxygen pressure and foot sense of touch. The foot ulcers are inspected for infection at every consultation, and a swab sample will be collected at enrollment. The size of the ulcers are measured and photographed each time. The investigators will count how many foot ulcers that are completely healed during the test period and measure the sizes of the remaining foot ulcers. The patients are asked to evaluate pain related to the foot ulcer. Data concerning participants' co morbidities and use of analgesic drugs are obtained from the patient journal and by patient interview.

Significance:

ESWT should be considered a supplement to existing clinical guidelines in wound management if shown to effectively help healing of diabetic foot ulcers. Improved healing should reduce the heavy workload on care and treatment regarding to these wounds. Hopefully, the frequency of amputations among diabetic patients will decline by implementing new treatment options for the diabetic foot.

DETAILED DESCRIPTION:
[Introduction]

It is estimated that 5.5 % of the Danish population suffers from diabetes - corresponding to more than 320.000 persons. Among Danish diabetic patients the yearly incidence of foot ulcers is higher than 3.000 and the prevalence higher than 22.000. Diabetics have a lifetime risk of foot ulcers of 15 %.

Amputation is a possible consequence to having a diabetic foot ulcer. A 19-year follow-up study performed on newly diagnosed diabetics shows an incidence of amputation of 400 per 100.000 patient years.

Economical costs associated with a diabetic foot ulcer vary with the severity and treatment of the ulcer. In Denmark costs including hospitalized treatment, outpatient treatment, homecare and other social services have been calculated to (written in Danish kroner 2009):

* Healed foot ulcer without ischemia: 152.800
* Healed foot ulcer with ischemia: 252. 800
* Foot ulcer with minor amputation: 407.900
* Foot ulcer with major amputation: 597.300

Groups including foot ulcers with minor or major amputation comprise 5 % of the total number of diabetic foot ulcers (corresponding to 150 amputations per year). Total costs of diabetic foot ulcers are 793 million Danish kroner.

Foot ulcers reduce the patients' mobility and their quality of life. Amputation is among the most feared complications to diabetes and it affects patients' quality of life as much as heart failure and cerebral stroke.

The treatment of diabetic foot ulcers is in several places of Denmark taken care of by multidisciplinary teams. Thus metabolic control, wound debridement, vascular surgery, treatment of infections, pain relief, occupational therapy etc. is taken care of in one specialized hospital unit. Parallel to a reorganization of the Danish health system 2000 - 2011 there was a significant decline in diabetic major amputations. However, no decline has been seen in the group of minor amputations and it may be that patients are now identified earlier for amputation thereby avoiding major amputations. Conclusively, a number of diabetic ulcer patients still cannot be offered any other treatment than amputation.

It is important to develop supplementing treatment options for the worst cases of diabetic foot ulcers. The goal is that ulcer healing is optimized and fewer patients are amputated.

In the field of diabetic foot ulcers a substantial amount of research is going on trying to develop existing methods of treatment and finding new therapeutic techniques. Extracorporeal shockwave therapy (ESWT) is a promising new option for ulcer treatment. ESWT has long been known in kidney stone treatment, and more recently ESWT has been established as treatment to regional pain disorders (such as plantar fasciitis of the heel and lateral epicondylitis of the elbow) and non-union of long bone fractures. Furthermore, ischemic heart disease and Peyronies disease have been treated with ESWT. Some studies show positive results when treating foot ulcers with ESWT.

In physics, shockwaves are high fluctuations of acoustical energy. When applied to a tissue shockwaves may stimulate an anabolic cellular response, increased blood perfusion and neo-angiogenesis. Shockwaves may furthermore promote anti-inflammatory effects and pain regulation. On a molecular scale upregulation of TGF-beta1, VEGF, FGF-2 signaling together with increased levels of NO and substance P in the tissue is seen following ESWT. During wound healing NO has been shown to induce IGF release through NF-kappaB pathway. Regarding to anti-inflammatory effects, ESWT reduces the cellular expression of metalloproteases and interleukins.

Clinical studies testing foot ulcer ESWT have not shown any significant side effects to shockwave treatment. These studies conclude that ESWT is safe to use.

----------------------------------------------------------------------------------------------------------------

[Purpose]

The investigators want to test if low-energy ESWT can help healing of complex diabetic foot ulcers. The effect of ESWT will be evaluated by measuring wound sizes and numbers of total healing, perception of pain using visual analog scale. Measures of cutaneous oxygen tension and foot sense of feeling will be included as well.

----------------------------------------------------------------------------------------------------------------

[Hypothesis]

ESWT improves diabetic patients' healing of chronic foot ulcers. In this study the investigators expect to see a faster wound area reduction among patients treated with ESWT compared to control group only receiving treatment according to current clinical guidelines.

Primary outcome measure for ESWT is

* Shorter time wound healing

Secondary outcome measures for ESWT are

* Pain reduction
* Increased perfusion
* No side effects

[Method]

Recruitment of patients: 6 months consecutive identification and inclusion of patients in Wound Clinic, Department of Plastic Surgery OUH. Every year approximately 400 patients with new ulcers are referred to the clinic. Patients who are either newly referred or in advance related to the clinic can be offered participation.

Randomization: Participants will be randomized to either intervention group or control group using a computer-generated table indicating allocation.

Intervention group: ESWT as a supplement to treatment following current clinical guidelines.

Control group: Ulcer treatment following clinical guidelines.

ESWT: A total of 6 times treatment over a 3 week period. Intervals between ESWT will be 3 - 4 days. ESWT will be carried out using the DUOLITH SD1 T-Top shockwave device, STORZ MEDICAL AG. The device is CE mark registered for ESWT use.

Description of intervention course: Participants in this group will have 8 consultations in a 7 week period. 6 times ESWT followed by 2 times follow-up respectively 2 and 4 weeks after last ESWT.

Description of control course: Participants in this group will have 4 consultations in a 7 week period. First consultation by enrollment. Second, third, and fourth consultations respectively 3, 5, and 7 weeks after enrollment. These four consultations corresponds to intervention group consultation number 1, 6, 7, and 8.

Baseline data: By the first consultation participants will be characterized in regard to the following variables:

* Sex
* Age
* Comorbidity (quantified using Charlson Index)
* Medical treatment: antidiabetics, analgesics (relevant drugs are NSAIDs, neuroleptics and opioids), antihypertensives, statins / cholesterol lowering drugs
* Smoking habits and alcohol consumption
* Body Mass Index
* Marital status, educational level and type of profession
* Classification of foot ulcer using University of Texas Wound Score
* Biochemistry: HbA1c, CRP, leukocytes, s-Na, s-K, s-creatinine, s-alkaline phosphatase, s-lactate dehydrogenase, s-cholesterol levels
* Bacterial colonization of the ulcer

Biochemical parameters and medical treatment data will be obtained from the patient records. New blood samples will be taken if the patient records do not include relevant test results - furthermore results must not be more than 2 months old.

Patients enrolled in the study will have access to all usually offered ulcer treatment. Information about other treatment modalities and frequencies will be obtained from participants patient records and patient interviews.

----------------------------------------------------------------------------------------------------------------

[Data handling]

Data will be noted in the REDCap online system. Data will be stored until study end. Analysis will be carried out using Stata software.

The study uses only one data collector who will also enter data in REDCap. However, if data are not available or missing, the specific measurements will be excluded from analysis. Missing data will be reported with published study results.

----------------------------------------------------------------------------------------------------------------

[Statistics]

Average percentage reduction of ulcer area is the study's primary end-point. If data are normally distributed (determined by probit or logit plot) statistical analysis can be performed using Student's t-test. Non-normally distributed data can be analyzed using transformation of data or non-parametric statistics (Wilcoxon rank sum test or Mann-Whitney U-test). Other numerical data (cutaneous oxygen tension, pain scoring, use of analgesics) can be statistically evaluated in the same manner as ulcer area reduction.

Complete ulcer healing is regarded as binary end-point data. Healing proportions will be calculated and compared between intervention group and control group - risk ratio and confidence intervals will be determined. Significance of data will be tested using Pearson's chi-squared test (alternatively Fisher's exact test if data material is small / does not fit chi-test). Sense of touch data will be evaluated in the same way.

Comparison of patient's quality of life in intervention group and control group is based on average questionnaire scores.

----------------------------------------------------------------------------------------------------------------

[Study power]

This study should be considered a pilot study. Earlier studies investigating ESWT ulcer treatment focus on study populations which are different from ours. The investigators consider our design to be unique since the investigators have not been able to identify earlier studies using a standard care control group to compare against intervention with 6 times ESWT in 3 weeks.

----------------------------------------------------------------------------------------------------------------

[Project feasibility]

The project is carried out as an undergraduate research year in the period 1/9-2014 - 1/9-2015. Medical student Sune Møller Jeppesen is accepted as an undergraduate student from the Faculty of Health Science, University of Southern Denmark. The undergraduate student works under guidance from main supervisor Lars Lund, professor, MD, DMSci. Knud Bonnet Yderstræde, MD, PhD, and Benjamin Schnack Rasmussen, MD, PhD-student, are co-supervisors for the project. Primarily, the undergraduate student's work will involve ESWT consultations and data collection. The student will be trained in relevant techniques needed for measuring ESWT effects.

Office facilities are available for the undergraduate student at the Department of Urology. Consultation room and devices for clinical measurements are available at the Wound Clinic, Department of Plastic Surgery OUH. Shockwave device will be purchased (see budget information).

The project will be registered to relevant authorities including the Danish Data Protection Agency and the Committee for Health Research Ethics, Denmark.

----------------------------------------------------------------------------------------------------------------

[Publication]

Trial results will be applied for publishing in an international scientific journal. Furthermore results will be presented at science conferences within the fields of interest.

----------------------------------------------------------------------------------------------------------------

[Economy]

The investigators seek research funding from private and public organizations. The investigators apply for 120.000 Danish kroner (DKK) to cover 12 months undergraduate student salary and 371.125 DKK for shockwave device purchase. Costs related to office facilities are 14.500 DKK. Project overhead is 3 % of total costs. Total project costs are 520.794 DKK.

----------------------------------------------------------------------------------------------------------------

[Significance of the project]

The project aims to evaluate healing effects of ESWT. If ESWT effectively can improve healing of complicated diabetic foot ulcers, ESWT should be considered for implementation in ulcer treatment clinical guidelines. Better ulcer healing can potentially improve patient's quality of life and decrease the number of diabetic patients who are being amputated (or at least postpone amputations). Later, research may be carried out to refine ulcer ESWT.

Proven ulcer healing effects of ESWT may also inspire future studies to test ESWT effects in the context of other clinical conditions. Possibly ESWT can be used in several settings where regenerative and anti-inflammatory effects are wanted.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving care and treatment in OUH Wound Clinic (Odense University Hospital, Denmark) with a diabetic foot ulcer.
* Wagner groups 1 and 2 (Wagner Ulcer Classification System)

Exclusion Criteria:

* Patients with an ulcer duration of less than 2 months
* Ulcer area less than 0,5 x 0,5 cm (or less than 0,25 cm2)
* Patients who have had vascular surgery performed within the past 2 months
* Patients who cannot give informed consent
* Patients who do not read or speak danish
* Wagner groups 3 and 4 (Wagner Ulcer Classification System)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Ulcer area | 49 days after enrollment
  We will use digital photos to determine 49 days ulcer area and compare to trial entry.

SECONDARY OUTCOMES:
Ulcer area (only intervention group) | 3-4 days after enrollment
  We will use digital photos to determine 3-4 days ulcer area and compare to trial entry.
Ulcer area (only intervention group) | 6-7 days after enrollment
  We will use digital photos to determine 6-7 days ulcer area and compare to trial entry.
Ulcer area (only intervention group) | 10-11 days after enrollment
  We will use digital photos to determine 10-11 days ulcer area and compare to trial entry.
Ulcer area (only intervention group) | 13-14 days after enrollment
  We will use digital photos to determine 13-14 days ulcer area and compare to trial entry.
Ulcer area (only intervention group) | 17-18 days after enrollment
  We will use digital photos to determine 17-18 days ulcer area and compare to trial entry.
Oxygen tension | 21 days after enrollment
  Cutaneous oxygen tension around ulcer
Oxygen tension | 35 days after enrollment
  Cutaneous oxygen tension around ulcer
Oxygen tension | 49 days after enrollment
  Cutaneous oxygen tension around ulcer
Pain | 21 days after enrollment
  Pain regarding to the ulcer will be assessed using Visual Analog Scale (VAS)
Pain | 35 days after enrollment
  Pain regarding to the ulcer will be assessed using Visual Analog Scale (VAS)
Pain | 49 days after enrollment
  Pain regarding to the ulcer will be assessed using Visual Analog Scale (VAS)
Side effects | 21 days after enrollment
  Side effects will be recorded by case history and clinical examination
Side effects | 35 days after enrollment
  Side effects will be recorded by case history and clinical examination
Side effects | 49 days after enrollment
  Side effects will be recorded by case history and clinical examination
Monofilament test | 21 days after enrollment
  Skin sensitivity on the foot will be tested by performing standardized monofilament test. Binary outcome measure.
Monofilament test | 35 days after enrollment
  Skin sensitivity on the foot will be tested by performing standardized monofilament test. Binary outcome measure.
Monofilament test | 49 days after enrollment
  Skin sensitivity on the foot will be tested by performing standardized monofilament test. Binary outcome measure.
Use of analgetics | 21 days after enrollment
  Participants use of analgetics will be recorded. Type and dosis will be noted.
Use of analgetics | 35 days after enrollment
  Participants use of analgetics will be recorded. Type and dosis will be noted.
Use of analgetics | 49 days after enrollment
  Participants use of analgetics will be recorded. Type and dosis will be noted.
Complete ulcer healing | 21 days after enrollment
  If ulcer is completely healed, this including time to event will be noted
Complete ulcer healing | 35 days after enrollment
  If ulcer is completely healed, this including time to event will be noted
Complete ulcer healing | 49 days after enrollment
  If ulcer is completely healed, this including time to event will be noted
Ulcer area | 21 days after enrollment
  We will use digital photos to determine 21 days ulcer area and compare to trial entry.
Ulcer area | 35 days after enrollment
  We will use digital photos to determine 21 days ulcer area and compare to trial entry.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Lund, Professor, Study Director — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

REFERENCES:
- [Background] Bruun C, Siersma V, Guassora AD, Holstein P, de Fine Olivarius N. Amputations and foot ulcers in patients newly diagnosed with type 2 diabetes mellitus and observed for 19 years. The role of age, gender and co-morbidity. Diabet Med. 2013 Aug;30(8):964-72. doi: 10.1111/dme.12196. Epub 2013 Apr 26. PMID 23617411
- [Background] Siersma V, Thorsen H, Holstein PE, Kars M, Apelqvist J, Jude EB, Piaggesi A, Bakker K, Edmonds M, Jirkovska A, Mauricio D, Ragnarson Tennvall G, Reike H, Spraul M, Uccioli L, Urbancic V, van Acker K, van Baal J, Schaper NC. Importance of factors determining the low health-related quality of life in people presenting with a diabetic foot ulcer: the Eurodiale study. Diabet Med. 2013 Nov;30(11):1382-7. doi: 10.1111/dme.12254. Epub 2013 Jul 15. PMID 23758490
- [Background] Vileikyte L. Psychosocial and behavioral aspects of diabetic foot lesions. Curr Diab Rep. 2008 Apr;8(2):119-25. doi: 10.1007/s11892-008-0022-1. PMID 18445354
- [Background] Goodridge D, Trepman E, Embil JM. Health-related quality of life in diabetic patients with foot ulcers: literature review. J Wound Ostomy Continence Nurs. 2005 Nov-Dec;32(6):368-77. doi: 10.1097/00152192-200511000-00007. PMID 16301902
- [Background] Alva M, Gray A, Mihaylova B, Clarke P. The effect of diabetes complications on health-related quality of life: the importance of longitudinal data to address patient heterogeneity. Health Econ. 2014 Apr;23(4):487-500. doi: 10.1002/hec.2930. Epub 2013 Jul 11. PMID 23847044
- [Background] Hirai FE, Tielsch JM, Klein BE, Klein R. Ten-year change in self-rated quality of life in a type 1 diabetes population: Wisconsin Epidemiologic Study of Diabetic Retinopathy. Qual Life Res. 2013 Aug;22(6):1245-53. doi: 10.1007/s11136-012-0245-0. Epub 2012 Aug 8. PMID 22872499
- [Background] Jorgensen ME, Almdal TP, Faerch K. Reduced incidence of lower-extremity amputations in a Danish diabetes population from 2000 to 2011. Diabet Med. 2014 Apr;31(4):443-7. doi: 10.1111/dme.12320. Epub 2013 Oct 21. PMID 24111834
- [Background] Game FL, Hinchliffe RJ, Apelqvist J, Armstrong DG, Bakker K, Hartemann A, Londahl M, Price PE, Jeffcoate WJ. A systematic review of interventions to enhance the healing of chronic ulcers of the foot in diabetes. Diabetes Metab Res Rev. 2012 Feb;28 Suppl 1:119-41. doi: 10.1002/dmrr.2246. PMID 22271737
- [Background] Gottrup F, Apelqvist J. Present and new techniques and devices in the treatment of DFU: a critical review of evidence. Diabetes Metab Res Rev. 2012 Feb;28 Suppl 1:64-71. doi: 10.1002/dmrr.2242. PMID 22271726
- [Background] Wang CJ. Extracorporeal shockwave therapy in musculoskeletal disorders. J Orthop Surg Res. 2012 Mar 20;7:11. doi: 10.1186/1749-799X-7-11. PMID 22433113
- [Background] Zimpfer D, Aharinejad S, Holfeld J, Thomas A, Dumfarth J, Rosenhek R, Czerny M, Schaden W, Gmeiner M, Wolner E, Grimm M. Direct epicardial shock wave therapy improves ventricular function and induces angiogenesis in ischemic heart failure. J Thorac Cardiovasc Surg. 2009 Apr;137(4):963-70. doi: 10.1016/j.jtcvs.2008.11.006. PMID 19327525
- [Background] Kiyota H, Ohishi Y, Asano K, Hasegawa N, Madarame J, Miki K, Kato N, Kimura T, Ishiyama T, Maeda S, Shimomura T, Shiono Y, Miki J. Extracorporeal shock wave treatment for Peyronie's disease using EDAP LT-02; preliminary results. Int J Urol. 2002 Feb;9(2):110-3. doi: 10.1046/j.1442-2042.2002.00430.x. No abstract available. PMID 12033197
- [Background] Schaden W, Thiele R, Kolpl C, Pusch M, Nissan A, Attinger CE, Maniscalco-Theberge ME, Peoples GE, Elster EA, Stojadinovic A. Shock wave therapy for acute and chronic soft tissue wounds: a feasibility study. J Surg Res. 2007 Nov;143(1):1-12. doi: 10.1016/j.jss.2007.01.009. Epub 2007 Sep 27. PMID 17904157
- [Background] Saggini R, Figus A, Troccola A, Cocco V, Saggini A, Scuderi N. Extracorporeal shock wave therapy for management of chronic ulcers in the lower extremities. Ultrasound Med Biol. 2008 Aug;34(8):1261-71. doi: 10.1016/j.ultrasmedbio.2008.01.010. Epub 2008 Apr 18. PMID 18394777
- [Background] Wang CJ, Kuo YR, Wu RW, Liu RT, Hsu CS, Wang FS, Yang KD. Extracorporeal shockwave treatment for chronic diabetic foot ulcers. J Surg Res. 2009 Mar;152(1):96-103. doi: 10.1016/j.jss.2008.01.026. Epub 2008 Mar 7. PMID 18619622
- [Background] Moretti B, Notarnicola A, Maggio G, Moretti L, Pascone M, Tafuri S, Patella V. The management of neuropathic ulcers of the foot in diabetes by shock wave therapy. BMC Musculoskelet Disord. 2009 May 27;10:54. doi: 10.1186/1471-2474-10-54. PMID 19473538
- [Background] Wang CJ, Wu RW, Yang YJ. Treatment of diabetic foot ulcers: a comparative study of extracorporeal shockwave therapy and hyperbaric oxygen therapy. Diabetes Res Clin Pract. 2011 May;92(2):187-93. doi: 10.1016/j.diabres.2011.01.019. Epub 2011 Apr 6. PMID 21310502
- [Background] Romeo P, Lavanga V, Pagani D, Sansone V. Extracorporeal shock wave therapy in musculoskeletal disorders: a review. Med Princ Pract. 2014;23(1):7-13. doi: 10.1159/000355472. Epub 2013 Nov 5. PMID 24217134
- [Background] Frairia R, Berta L. Biological effects of extracorporeal shock waves on fibroblasts. A review. Muscles Ligaments Tendons J. 2012 Apr 1;1(4):138-47. Print 2011 Oct. PMID 23738262
- [Background] Notarnicola A, Moretti B. The biological effects of extracorporeal shock wave therapy (eswt) on tendon tissue. Muscles Ligaments Tendons J. 2012 Jun 17;2(1):33-7. Print 2012 Jan. PMID 23738271
- See also: Statens Serum Institut (SSI) is responsible for research-based health surveillance, rational use of IT in the Danish healthcare system and prevention and control of infectious diseases, biological threats and congenital disorders. — http://www.ssi.dk/Sundhedsdataogit/Sundhedsvaesenet%20i%20tal/Specifikke%20omraader/Diabetes.aspx